CLINICAL TRIAL: NCT04943549
Title: Erector Spinae Plane Block Impact on Quality of Recovery After Lumbar Spinal Decompression Surgery; a Comparative Study Between Addicts and Non-addicts
Brief Title: Erector Spinae Plane Block Impact on Quality of Recovery After Lumbar Spinal Decompression
Acronym: ESPB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Abdel Fatah, Lecturer, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5-5-2021
Record Dates: First submitted 2021-06-08; First posted 2021-06-29 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Pain
Keywords: Lumber surgery; Postoperative analgesia; Erector spinae pain block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Active Comparator): History of addiction.
  Interventions: Drug: Bupivacain
- Group (N) (Placebo Comparator): No history of addiction to any drug.
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — Patients will be placed in left lateral position. A low-frequency curved array ultrasound transducer will be used. The ultrasound transducer will be placed in a longitudinal orientation 2-3 cm lateral to the midline to identify the hyperechoic line of the transverse process. After identification of muscles superficial to the transverse process and local infiltration of anesthesia into the superficial tissues, a block needle will be inserted in a craniocaudal direction until contact will be achieved with the transverse process where the tip will lay in the interfascial plane below the erector spinae muscle. A small bolus of local anaesthetic should be given through the block needle; the erector spinae muscle should be visualized, separating from the transverse process. A total of 20 mL bupivacaine 0.25% will be injected into the interfacial plane deep to the erector spinae muscle bilaterally. Forty minutes after the ESPB, the cutaneous sensory block will be assessed.

SUMMARY:
Erector spinae plane block (ESPB) as a new trunk fascia block technique was proposed in 2016. ESPB has aroused the interest of many nerve block experts. The benefits of ESPB are not yet demonstrated. The specific mechanism is still controversial. Some believe that ESPB can block the posterior root of the spinal nerve and produce part of the para-spinal block effect with the diffusion of the drug solution.

The present study will carried out to compare the performance of the erector spinae plane block combined with general anesthesia in addicts versus non addicts' patients regarding the local analgesic effect, recovery after surgery and side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male gender.
2. Age range of 18-60 years.
3. Scheduled for open lumbar decompression surgery.
4. A minimum of 1-year experience of drug consumption or having drug withdrawal symptoms when stopping for inclusion in the drug addicts group(according to the patient's statement and rapid opiate urine test).

Exclusion Criteria:

1. Hepatic or renal insufficiency.
2. Preoperative cognitive dysfunction or communication disorder.
3. Allergy to amide-type local anaesthetics.
4. Back puncture site infection.
5. Coagulation disorders.
6. Emergency surgery.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
The quality of recovery score (QoR-15) at 24th hour | at 24th hour
  This questionnaire covers a total of 15 questions under five clinical dimensions of health; physical comfort (five-item), emotional status (four-item), psychological support (two-item), physical independence (two-item) and pain (two-item). a numerical rating scale of 11 point for each question leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).

SECONDARY OUTCOMES:
Postoperative pain. | At half an hour, 2, 4, 8, 12, 24 hours.
  Postoperative pain assessed by VAS which scales from zero (no pain) to ten (unbearable pain).
  .
Intraoperative fentanyl dosage. | From the start of operation till its end up to 3 hours.
  Intraoperative fentanyl dosage (μg)
First-time morphine use. | In 24 hours
  First-time morphine use(in hours).
First time to ambulation after surgery. | In 24 hours
  First time to ambulation after surgery(in hours).
Length of hospital stay. | up to 3 days.
  It is the time of postoperative patient's stay in hospital till discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Banha Faculity of Medicine, Banhā, Elqalyoubea, Egypt